CLINICAL TRIAL: NCT05215925
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Safety of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) in Advanced nsqNSCLC Patients With High EGFR Expression
Brief Title: A Study to Evaluate the Efficacy and Safety of HLX07 in nsqNSCLC Patients With High EGFR Expression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-nsqNSCLC201
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-05

CONDITIONS: HLX07, nsqNSCLC, High EGFR Expression
MeSH Terms: interventions — HLX07

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: HLX07+carboplatin+pemetrexed
- B (Experimental)
  Interventions: Drug: HLX07+docetaxel
- C (Experimental)
  Interventions: Drug: HLX07

INTERVENTIONS:
Drug: HLX07+carboplatin+pemetrexed — HLX07 1500mg q3w+carboplatin+pemetrexed
  Other Names: Anti-EGFR Monoclonal Antibody
  Arms: A
Drug: HLX07+docetaxel — HLX07 1500mg q3w+docetaxel
  Arms: B
Drug: HLX07 — HLX07 1500mg q3w
  Arms: C

SUMMARY:
An Open-label, Multicenter , Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) in Combination with Chemotherapy or Monotherapy in Advanced Non-squamous Non-small Cell Lung Cancer (nsqNSCLC) Patients with High EGFR Expression

ELIGIBILITY:
Inclusion Criteria:

1. Age>=18Y
2. Good Organ Function
3. Expected survival time ≥ 3 months
4. Histologically confirmed, advanced/recurrent or metastatic nsqNSCLC
5. Measurable lesion according RECISTv1.1 by investigator
6. High EGFR expression H score ≥200
7. ECOG score 0-1

Exclusion Criteria:

1. Histologically, squamous NSCLC should be excluded. For tumors with adenocarcinoma and squamous carcinoma, if the adenoid component is dominant and the squamous component is < 5%, the patients meet the inclusion requirements.
2. Previous treatment with EGFR inhibitors
3. Symptomatic brain or meningeal metastases (unless the patient has been on > treatment for 3 months, has no evidence of progress on imaging within 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable).
4. Active clinical severe infection;
5. A history of other malignancies within 5 years, except for cured carcinoma in situ of the cervix or basal cell carcinoma of the skin,etal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the RECIST Version 1.1)
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (PFS) (assessed by IRRC and the investigator as per RECIST v1.1

SECONDARY OUTCOMES:
OS | from the date of first dose until the date of death from any cause，assessed up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China